CLINICAL TRIAL: NCT07317219
Title: Effects of a Single Dose of Ayahuasca or Esketamine on Body Image Perception in Women: a Randomized, Double-blind Study
Brief Title: Ayahuasca, Esketamine and Body Image Perception
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Rafael Guimarães dos Santos, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 83923024.0.0000.5440
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Healthy Women Volunteers
MeSH Terms: interventions — Esketamine; Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ayahuasca (Experimental): oral ayahuasca
  Interventions: Drug: Ayahuasca
- esketamine (Active Comparator): oral esketamine
  Interventions: Drug: Esketamine

INTERVENTIONS:
Drug: Ayahuasca — oral ayahuasca
  Other Names: aya
  Arms: ayahuasca
Drug: Esketamine — oral esketamine
  Other Names: ketamine
  Arms: esketamine

SUMMARY:
Double-blind, randomized trial comparing a single dose of oral ayahuasca or esketamine on women body perception.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers

Exclusion Criteria:

* psychiatric and other medical comorbidities

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — healthy women
Enrollment: 20 (Estimated)
Dates: Start 2025-12-20 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Body Shape Questionnaire | From enrollment to the end of treatment at 3 weeks
  higher scores mean a worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital das Clínicas da FMRP-USP, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No